CLINICAL TRIAL: NCT04809857
Title: The Effect of Plyometric Exercises on Muscle Strength in Premenopausal Women
Brief Title: Effect of Plyometric Exercises in Premenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Kübra Alpay, Lecturer of Pysiotherapy and Rehabilitation Department, Bezmialem Vakif University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Kubra2
Record Dates: First submitted 2021-02-17; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Premenopausal Women
Keywords: Plyometric exercise; Isokinetic; Muscle strength; Premenopause
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Plyometric Exercise Group (Experimental): Plyometric exercise training 3 days a week for 6 weeks
  Interventions: Other: Exercise
- Isokinetic Exercise Group (Active Comparator): Isokinetic exercise training 3 days a week for 6 weeks
  Interventions: Other: Exercise
- Control Group (No Intervention): no exercise intervention

INTERVENTIONS:
Other: Exercise
  Arms: Isokinetic Exercise Group; Plyometric Exercise Group

SUMMARY:
It was aimed to examine the effects of plyometric exercises on muscle strength in this study. 26 premenopausal women assigned to one of the three groups: Control Group (n=8), Plyometric Exercise Group (n=10) and Isokinetic Exercise Group (n=8). Muscle strength assessments, depression and anxiety inventories were performed baseline and after 6 weeks.

DETAILED DESCRIPTION:
Depending on various factors, bone mass begins to decrease with aging and this may lead to the osteoporosis. Physical activity and regular exercise provides an increase in bone mineral density (BMD). It is mentioned that there are relationships between muscle strength and BMD and also muscle strength has positive effects on BMD. In the literature it is showed that postmenopausal women with weaker trunk muscle strength could have risk of osteoporosis.

Plyometric exercises are used to increase muscle strength. Physiological basis of plyometric exercise consist of stretch-shortening cycle and thus it is effective in increasing the force. At the same time, plyometric exercises have positive effects on BMD because of weight bearing exercises.

The aim of this study was to investigate the effects of plyometric exercises on hip and trunk muscle strength in premenopausal women.

Participants and Study Design: Twenty six sedentary premenopausal women aged 35-50 years participated this study. Participants were assigned into three groups: Plyometric Exercise Group (PG; n=10), Isokinetic Exercise Group (IG; n=8), Control Group (CG; n=8). Participants were informed about the procedures of the study and signed a written voluntary consent form in accordance with the Declaration of Helsinki. The study protocol was approved by the Ethical Committee of the Istanbul University Medical Faculty. Measurements and training sessions were performed in the Istanbul University Medical Faculty Sport Medicine Department's Laboratory.

Measurements: Muscle strength was determined by using a Cybex Norm isokinetic dynamometer (Cybex Humac Norm, USA). Range of motion was set from 10 degree extension to 40 degree flexion. Isokinetic concentric contraction strength was measured at angular velocity of 60 degree per second and 90 degree per second. Subjects performed 3 trials trunk flexion and extension contractions at minimal exertion and 4 test repetitions at maximal trunk flexion and extension.

The hip abduction adduction isokinetic testing was performed in side lying position. Hip muscle strength was measured at angular velocity of 30 degree per second. Range of motion was set from 10 degree adduction to 40 degree abduction. Subjects performed 4 trials at minimal exertion and 4 test repetitions. Dominant leg values were analyzed for hip. All subjects performed warm-up and stretching exercises before testing.

Beck Depression Inventory (BDI) and State-Trait Anxiety Inventory (STAI) were used to asses depression and anxiety conditions.

Interventions: The training sessions were performed three days a week for six weeks. All exercise sessions were supervised by a physiotherapist.

Each session was consisted of warm-up, plyometric exercises and cool-down periods in PG. The warm-up and cool-down periods were performed by walking on the treadmill and lower extremity stretching exercises. The plyometric exercise training period involved vertical jumping, forward and back jumping and lateral jumping. After fifth session the number of repetitions were increased depending of toleration of participants. After tenth session step bench jumping exercise and after fifteenth session diagonal jumping exercise were added and study was completed in eighteen session.

In IG, isokinetic exercises were performed by using a Cybex Norm isokinetic dynamometer with an incorporated trunk flexion/extension unit in a standing position. Range of motion was set from 10 degree extension to 40 degree flexion. Each session was consisted warm-up, isokinetic exercises and cool-down periods. Warm-up and cool-down periods were consisted trunk exercise and stretching. Isokinetic exercises were performed 7 repetitions at angular velocity of 90 degree per second , 6 repetitions at angular velocity of 75 degree per second and 5 repetitions at angular velocity of 60 degree per second.

Participants in CG were assessed baseline and at sixth week.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women aged 35-50 years

Exclusion Criteria:

* to have cardiovascular, musculoskeletal and neurologic disease
* have been involved in exercise studies within the last 6 months
* to being receive hormone replacement therapy

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2007-02 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Isokinetic testing trunk flexion-extension | Six weeks
  changes trunk flexion and extension muscle strength from baseline at 6 weeks
Isokinetic testing hip abduction-adduction | Six weeks
  changes hip abduction and adduction muscle strength from baseline at 6 weeks

SECONDARY OUTCOMES:
Beck Depression Inventory | Six weeks
  changes inventory scores from baseline at 6 weeks
State Trait Anxiety Inventory | Six weeks
  changes inventory scores from baseline at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Safinaz Yildiz, Study Director — Istanbul University; Kubra Alpay, Principal Investigator — Bezmialem Vakif University; Turker Sahinkaya, Study Chair — Istanbul University

IPD SHARING:
Plan to Share IPD: No